CLINICAL TRIAL: NCT06381765
Title: Comparison of Deep Serratus Plane Block with Deep Serratus Plane Block+Pectointercostal Plane Block
Brief Title: Serratus Plane Block and Pectointercostal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Associate professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Serratus-Pectointercostal
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Serratus plane block (Active Comparator): Deep serratus plane block will perform with 20 ml 0,25 %bupivacaine at the midaxillary 5. rib, bilaterally
  Interventions: Procedure: ultrasound guided Serratus plane bock
- Serratus plane block+pectointercostal plane block (Active Comparator): deep serratus plane block (20 ml 0,25 %bupivacaine) at the midaxillary 5.th rib+ pectointercostal plane block (0,25% bupivacaine 15 ml) at 4-5.th intercostal space will perform bilaterally .
  Interventions: Procedure: ultrasound guided Serratus plane bock and pectointercostal block

INTERVENTIONS:
Procedure: ultrasound guided Serratus plane bock and pectointercostal block — ultrasound guided serratus plane block (20 ml 0,25 %bupivacaine) will perform at the midaxillary 5.th rib and pectointercostal plane block (0,25% bupivacaine 15 ml) will perform at 4-5.th intercostal space. Both 2 blocks will perform bilaterally
  Arms: Serratus plane block+pectointercostal plane block
Procedure: ultrasound guided Serratus plane bock — ultrasound guided serratus plane block (20 ml 0,25 %bupivacaine) will perform at the midaxillary 5.th rib to the all patients
  Arms: Serratus plane block

SUMMARY:
ASA I-II female patients aged over 18 who will undergoing breast reduction surgery will recruit to the study. Patients will divide into 2 groups. Deep serratus plane block will perform with 0,25 %bupivacaine 20 ml at the midaxillary 5. rib, bilaterally for Group I. At Group II, deep serratus plane block ( 0,25 %bupivacaine 20 ml) at the midaxillary 5.th rib+ pectointercostal plane block (0,25% bupivacaine 15 ml) at 4-5.th intercostal space will perform bilaterally . General anesthesia with sevoflurane and remifentanil will perform to the all patients. Postoperative pain scores, morphine consumption and complications will record till the 24.th hours.

DETAILED DESCRIPTION:
ASA I-II female patients aged over 18 who will undergoing breast reduction surgery will recruit to the study. General anesthesia with sevoflurane and remifentanil will perform to the all patients. Patients will divide into 2 groups. Serratus plane block for group I and serratus plane block+pectointercostal block for Group II will perform bilaterally. Ultrasound guided deep serratus plane block will perform with 0,25% bupivacaine 20 ml at the midaxillary 5. rib, for Group I. At Group II, ultrasound guided deep serratus plane block ( 0,25 %bupivacaine 20 ml) at the midaxillary 5.th rib+ pectointercostal plane block (0,25% bupivacaine 15 ml) at 4-5.th intercostal space will perform bilaterally. Patient controlled analgesia will perform with Morphine ( 1 mg bolus+ 10 min lockout+4 hours limit 10 mg) at postoperative period. Patients will evaluate with visual analogue scale (VAS) for postoperative pain scores till the first 24.th hours. Postoperative pain scores (VAS), morphine consumption and complications will record till the 24.th hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Female
* who will undergoing Breast reduction surgery

Exclusion Criteria:

* ASA III and over patients
* who reject to join the study
* male gender

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-65 aged females.
Enrollment: 60 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
postoperative morphine consumption | All the patients will follow till the postoperative 24.th hours and totally morphine consumption will record postoperative 24.th hours.
  Patient controlled analgesia with morphine will perform to the all patients and morphine consumption will calculate and record till the end of 24.th hours.
postoperative visual analog scale scores | VAS scores will record at the first postoperative 24.th hours
  All the patients will evaluate with visual analog scale scores (VAS) at the first postoperative 24.th hours period. VAS scores will define between 0-10 scores. 0 score means lowest pain score and 10 means the worst pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Biricik, Principal Investigator — çukurova university faculty of medicine
Locations (1):
- Çukurova University Faculty of Medicine, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No